CLINICAL TRIAL: NCT00724607
Title: Validation of Brief Objective Neurobehavioral Detectors of Mild TBI
Brief Title: Brain Injury Outcomes (BIO) Study
Acronym: BIO
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oak Ridge National Laboratory (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: SHP 08-167; 01133 (Other: IRB)
Record Dates: First submitted 2008-07-23; First posted 2008-07-29 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Brain Concussion; Posttraumatic Stress Disorder; Dementia
Keywords: Concussion, traumatic brain injury; Screening; neuroimaging; Posttraumatic stress disorder; Longitudinal studies
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Dementia; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — We are not collecting tissue samples at this time due to staffing shortages in our research service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- TBI (Case) Group: Members of the TBI group have sustained a TBI in accordance with inclusion/exclusion criteria. However, the investigative staff administering, scoring, analyzing and interpreting the data will be blinded to the group status of the participant.
- Non-TBI (Control) Group: Members of the Non-TBI group have not sustained a TBI and are in accordance with other provisions of the inclusion/exclusion criteria. However, the investigative staff administering, scoring, analyzing and interpreting the data will be blinded to the group status of the participant. This longitudinal study will utilize a control group to account for normal aging and other control factors.
- Non-TBI Non-deployed (Control) Group: Members of the Non-TBI Non-Deployed group have neither sustained a TBI nor have been deployed but are in accordance with other provisions of the inclusion/exclusion criteria. However, the investigative staff administering, scoring, analyzing and interpreting the data will be blinded to the group status of the participant. This longitudinal study will utilize this Non-deployed control group to account for deployment-specific factors.

SUMMARY:
Many active duty military, national guard, and reserves personnel who served in the recent conflicts in Afghanistan and Iraq were exposed to blasts and other mechanisms of traumatic brain injury (TBI).1,2 Although physical trauma is not unexpected during war fighting, survival after head injury, particularly blast-related, has become a common occurrence only in recent decades. As such, the associated cerebral damage is less well studied and understood, particularly over the long term.

The Brain Injury Outcomes (BIO) is a longitudinal study with the short-term objective of better characterizing multi-modal outcomes in individuals who have sustained a brain injury using a systems medicine approach. Long-term aims include monitoring participants for signs of emerging symptoms or age-related vulnerabilities. Identification of abnormality profiles for multiple severity levels of brain injury (from any source, including blast and non-blast) reflects a second long-range goal. Third, the investigators will examine and compare physiology between Veterans who have sustained a Mild Traumatic Brain Injury (mTBI) with and without persisting symptoms and various co-morbidities including posttraumatic stress disorder (PTSD) and depression. A control group of Veterans who have not sustained a TBI will also be recruited for comparison. Fourth, the investigators intend to facilitate the clinical use of advanced methodologies, such as brain imaging measures, with the brain injured (and other populations). Finally, the investigators will assess methods of analysis, separately and in combination through integration, for multi-modal data in search of diagnostic profiles. Increased knowledge of injury patterns and the trajectory associated with brain injury could contribute to better methods of diagnosis, monitoring and, perhaps, treatment.

This investigation has spawned several sub-studies, one of which was the Validation of Brief Objective Neurobehavioral Detectors (BOND) of Mild TBI, which continues. The investigators have collaborated with Harvard/Boston Children's Hospital in the Angiogenic Signaling Signatures Identified in Stress and Trauma (ASSIST) sub-study. Oak Ridge National Laboratory (ORNL) will assist in integrating BIO Study multi-modal data. Investigators at Johns Hopkins School of Medicine collaborate with neuroimaging sequences and methods.

DETAILED DESCRIPTION:
This study was previously paused due to the pandemic.

Many active duty military, national guard, and reserves personnel who served in the recent conflicts in Afghanistan and Iraq were exposed to blasts and other mechanisms of traumatic brain injury (TBI).1,2 Although physical trauma is not unexpected during war fighting, survival after head injury, particularly blast-related, has become a common occurrence only in recent decades. As such, the associated cerebral damage is less well studied and understood, particularly over the long term.

The Brain Injury Outcomes (BIO) is a longitudinal study with the short-term objective of better characterizing multi-modal outcomes in individuals who have sustained a brain injury using a systems medicine approach. Long-term aims include monitoring participants for signs of emerging symptoms or age-related vulnerabilities. Identification of abnormality profiles for multiple severity levels of brain injury (from any source, including blast and non-blast) reflects a second long-range goal. Third, the investigators will examine and compare physiology between Veterans who have sustained a Mild Traumatic Brain Injury (mTBI) with and without persisting symptoms and various co-morbidities including posttraumatic stress disorder (PTSD) and depression. A control group of Veterans who have not sustained a TBI will also be recruited for comparison. Fourth, the investigators intend to facilitate the clinical use of advanced methodologies, such as brain imaging measures, with the brain injured (and other populations). Finally, the investigators will assess methods of analysis, separately and in combination through integration, for multi-modal data in search of diagnostic profiles. Increased knowledge of injury patterns and the trajectory associated with brain injury could contribute to better methods of diagnosis, monitoring and, perhaps, treatment.

This investigation has spawned several sub-studies, one of which was the Validation of Brief Objective Neurobehavioral Detectors (BOND) of Mild TBI, which continues. The investigators have collaborated with Harvard/Boston Children's Hospital in the Angiogenic Signaling Signatures Identified in Stress and Trauma (ASSIST) sub-study. Oak Ridge National Laboratory (ORNL) will assist in integrating BIO Study multi-modal data. Investigators at Johns Hopkins School of Medicine collaborate with neuroimaging sequences and methods.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for TBI Group (Case Group):

TBI group Veterans must:

* be enrolled at the Washington, DC VA Medical Center
* be an Operation Enduring Freedom (OEF)/ Operation Iraqi Freedom (OIF)/OND Veteran
* be between the ages of 18 and 59, inclusive
* have at least 10 years of education
* be able to fit into scanner (i.e., weigh less than 400 pounds)
* have a brain injury (based upon VHA criteria)
* be at least one year post-injury

Inclusion criteria for NonTBI Group (Control Group):

NonTBI group Veterans must:

* be enrolled at the Washington, DC VAMC
* have been active duty (whether deployed or not) during OEF and/or OIF and/or OND
* be between the ages of 18 and 59, inclusive
* have at least 10 years of education

Exclusion Criteria:

Exclusion Criteria for both the Case and Control Groups:

Veterans must NOT:

* be colorblind or have any visual impairment that interferes with reading or writing
* have any upper extremity dysfunction that prevents the use of a pencil or computer mouse or keyboard
* meet criteria for substance dependence within 1 month of the evaluation
* have a current acute or unstable psychiatric condition
* have a current diagnosis (or symptoms consistent with) schizophrenic or bipolar disorders, or severe uni-polar depression
* be in significant pain during the evaluation (patient subjective report)
* have a diagnosis of diabetes (PET imaging considerations)
* have had or currently have any other injury, medical or neurological illness, or exposure that could potentially explain cognitive deficits (e.g., Central Nervous System disease, prior brain injury, seizure disorder, or HIV)
* be taking prescription drugs that significantly interfere with outcome measures
* have any devices or material implanted, embedded, or attached to the body containing ferrous material that interferes with MR imaging (i.e., pacemaker, shrapnel)
* Be a pregnant or lactating female (MRI considerations)
* Display behavior that would significantly interfere with validity of data collection or safety during study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: OEF/OIF/OND Veterans with and without mTBI and/or PTSD
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2008-05-06 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy (FA) | Alternating years
  In this longitudinal study with multiple measurement modalities (i.e., neuroimaging, neurologic exam, cognition, etc.), the primary outcome measures are from the neuroimaging modality, specifically, the diffusion tensor imaging (DTI) sequences. FA is one of the quantitative metrics yielded by the DTI sequence. FA is a ratio of the directional flows of water molecules within axonal bundles and is interpreted as a representation of the overall structural health of the bundle.

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Chapman, PsyD, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing via de-identified individual participant databases propels research efforts forward by allowing other qualified researchers to conduct subsequent studies more efficiently with less patient burden. However, the original consent forms for the BIO Study (began in 2008) did not specify such a sharing plan. As such all participants would have to be re-consented in order to pursue such a data sharing plan. The PI and Investigative Team are in favor of providing an option to participants so that they could choose whether or not they would want their de-identified data to be available for other researchers to utilize for future study.

REFERENCES:
- See also: PubMed Abstract — http://www.ncbi.nlm.nih.gov/pubmed/20599047